CLINICAL TRIAL: NCT03511755
Title: A 12-Week, Multicenter, Double-Blind, Controlled, Randomized Study Assessing Change in Psoriasis Severity and Level of Stress in Patients With Moderate to Severe Psoriasis Using Transdermal Electrical Neurosignaling (TEN)
Brief Title: 12-Week Study Assessing Change in Psoriasis Severity and Level of Stress Using TEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thync Global, Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THY-002
Record Dates: First submitted 2018-04-03; First posted 2018-04-30 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Psoriasis; Stress
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TEN 1-11 kHz (Experimental): Transdermal Electrical Neuromodulator (TEN) waveform pulsed biphasic current (1-11 kHz)
  Interventions: Device: Transdermal Electrical Neuromodulator (TEN)
- TEN 1-3 kHz (Active Comparator): Transdermal Electrical Neuromodulator (TEN) waveform pulsed biphasic current (1-3 kHz)
  Interventions: Device: Transdermal Electrical Neuromodulator (TEN)

INTERVENTIONS:
Device: Transdermal Electrical Neuromodulator (TEN) — Thync TEN is a portable, battery-powered, electrical neuromodulation device connected to single-use gel electrode pads that are applied to the base of the neck (C3 to C7).
  Other Names: Thync TEN

SUMMARY:
This is a 12-Week, multicenter, double-blind, controlled, randomized study assessing change in psoriasis severity and level of stress in patients with moderate to severe psoriasis treated with TEN. Psoriasis severity and stress levels will be measured at Weeks 0, 4, 8 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female of any race, 18 years of age or older.
* Moderate (>3 to <10% BSA) with a PASI of at least 6 and less than 12 or severe (≥10% BSA) plaque psoriasis with a minimal PASI score of 12.
* Subject diagnosed with psoriasis at least 6 months prior to entering the study.
* Subjects who have received treatment in the past for psoriasis and are currently untreated or subjects who are on stable treatment for psoriasis that is expected to remain unchanged throughout the entire duration.
* Subjects who have not received psoriasis treatments in the past should be stable in their disease for the last 4 weeks.

Exclusion Criteria:

* Guttate, erythrodermic, or pustular psoriasis subtypes.
* Evidence of skin conditions other than psoriasis that would interfere with study-related evaluations of psoriasis.
* Unstable psoriasis or unstable treatment of psoriasis over the entire duration of the study.
* Subjects with moderate psoriasis are not allowed to use concurrent systemic therapies for psoriasis (i.e., phototherapy, orals, biologics, etc.). Topical medications are allowed;
* Subjects with severe psoriasis are allowed to use any concurrent therapy for psoriasis, provided that disease state is stable for ≥2 months and they meet minimum PASI requirements.
* Cardiac pacemaker, implanted defibrillator, or other implanted metallic or electronic device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who reach PASI 50 (50% reduction in PASI score from Baseline) | Week 4, 8, and 12
  Standard Psoriasis Area and Severity Index (PASI) scoring system, which incorporates erythema, induration, and scale (0-4) weighted by percentage of body surface area involvement.
Proportion of subjects who reach PASI 75 (75% reduction in PASI score from Baseline) | Week 4, 8, and 12
  Standard Psoriasis Area and Severity Index (PASI) scoring system, which incorporates erythema, induration, and scale (0-4) weighted by percentage of body surface area involvement.

SECONDARY OUTCOMES:
PASI change from Baseline | Week 4, 8, and 12
  Standard Psoriasis Area and Severity Index (PASI) scoring system, which incorporates erythema, induration, and scale (0-4) weighted by percentage of body surface area involvement.
IGA change from Baseline | Week 4, 8, and 12
  Standard Investigator Global Assessment (IGA) scoring system, which incorporates plaque elevation, scaling and erythema on a score of 0-5 (clear to very severe) averaged over all lesions.
IGA Responder Rate | Week 4, 8, and 12
  Proportion of Subjects with a Standard Investigator Global Assessment (IGA) score of 0 or 1. IGA incorporates plaque elevation, scaling and erythema on a score of 0-5 (clear to very severe) averaged over all lesions.
DLQI change from Baseline | Week 4, 8, and 12
  Dermatology Life Quality Index 10-item self-reported survey, to addresses feelings, daily activities, leisure, work, school, personal relationships, and treatment. Each question item is worth 3 points (total maximum score of 30), with higher score representing greater QoL impairment.
PQOL-12 change from Baseline | Week 4, 8, and 12
  Psoriasis Quality of Life - 12 Item psoriasis-specific validated Patient Reported Outcome questionnaire, developed as part of the Koo-Menter Psoriasis Index (KMPI) in 2005, a tool to determine whether a patient with moderate to severe psoriasis is a candidate for more aggressive treatments beyond topical therapies.
HADS change from Baseline | Week 4, 8, and 12
  Hospital Anxiety and Depression Scale self-rated 14-item questionnaire, with seven questions related to depression (HADS-D) and seven to anxiety (HADS-A). Scoring is interpreted as follows: 0-7 points is defined as no symptoms, 8-10 points are mild symptoms, 11-14 points signify moderate symptoms, and severe symptoms are defined as having greater than 15 points. Depression and anxiety states are diagnosed when HADS-D and HADS-A scores are greater than 8 points, respectively.
QVAS change from Baseline | Week 4, 8, and 12
  Stress Level Quantified Visual Analogue Scale (QVAS) subjective measure of level of stress using an 11-point scale (0-10)
Pruritus NRS change from Baseline | Week 4, 8, and 12
  Pruritus Numerical Rating 11-point Scale (0-10) to assess subjective maximum itch intensity in the previous 24 hours

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Site 1, Fremont, California
  - Site 3, San Diego, California
  - Site 2, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No